CLINICAL TRIAL: NCT01489150
Title: Use of EtCO2 and Prolonged Expiratory Maneuvers as a PaCO2 Predictor in Cases of Acute Hypercapnic Respiratory Failure
Brief Title: Use of EtCO2 as a PaCO2 Predictor Under Non Invasive Ventilation (NIV) in Cases of Acute Hypercapnic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Philippe Jolliet, Principal investigator, University of Lausanne Hospitals
Other Study IDs: EtCO2-NIV
Record Dates: First submitted 2011-12-02; First posted 2011-12-09 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Hypercapnic Respiratory Failure
Keywords: Acute respiratory failure; Hypercapnia; Non invasive ventilation; End-tidal CO2
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients treated by Non invasive ventilation (NIV) due to acute hypercapnic respiratory failure, the interest of using the End-tidal Co2 measurement device "Capnostream" to evaluate PaCo2 and PaCo2 variations over time will be evaluated. Measurements will be done under normal expiration and under prolonged active and passive expiration maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient equipped with arterial line
* NIV requirement
* Hypercapnia: PaCO2 > 45mmhg

Exclusion Criteria:

* Severe hemodynamic instability
* Severe psychiatric disorders
* nasal lesions
* denied consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients equipped with arterial line requiring non invasive ventilation because of acute hypercapnic respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Comparison between EtCO2,PaCO2 and PaCO2 variation under NIV during both spontaneous expiration and prolonged expiration | Sixty minutes
  Comparison between EtCO2,PaCO2 and PaCO2 variation under NIV during both spontaneous expiration and prolonged expiration

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jolliet, Professor, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Intensive care and burn unit, University Hospital of Lausanne, Lausanne, Switzerland

REFERENCES:
- [Derived] Piquilloud L, Thevoz D, Jolliet P, Revelly JP. End-tidal carbon dioxide monitoring using a naso-buccal sensor is not appropriate to monitor capnia during non-invasive ventilation. Ann Intensive Care. 2015 Feb 12;5:2. doi: 10.1186/s13613-014-0042-8. eCollection 2015. PMID 25852962